CLINICAL TRIAL: NCT03051425
Title: Immune Benefits of Consumption of Dairy Yogurt Containing Functional Probiotics Among Individuals Over 60 Years Old
Brief Title: Immune Benefits of Consumption of Dairy Yogurt in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CI_immune
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Immune Deficiency
Keywords: Probiotics; Immune function; Natural killer cell activity; Interleukin-12; Interferon-gamma; Immunoglobulin
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Probiotic yogurt supplementation
  Interventions: Dietary Supplement: Probiotic yogurt
- Placebo group (Placebo Comparator): Placebo supplementation
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic yogurt — 120 mL of Yogurt containing Lactobacillus delbrueckii subsp. bulgaricus, Streptococcus thermophilus, Lactobacillus casei, Bifidobacterium animalis ssp. lactis, and Lactobacillus plantarum
  Arms: Test group
Dietary Supplement: Placebo — 120 mL of low-fat milk
  Arms: Placebo group

SUMMARY:
To investigate the impact of consuming dairy yogurt on immun function including natural killer (NK) cell activity, circulating levels of cytokines, and immunoglobulin (Ig) in elderly.

DETAILED DESCRIPTION:
A randomized, open-labelled, placebo-controlled study was conducted on 200 nondiabetic, nonobese and elderly (≥60 years) subjects. Over a twelve-week period, the test group consumed one bottle (120 mL) of dairy yogurt each day, whereas the placebo group consumed same volume of low fat milk daily. NK cell activity (%) was measured based on the ratios of effector cells (E; peripheral blood mononuclear cells, PBMCs) from each participant to target cells (T; K562 cells) at E:T= 10:1, 5:1, 2.5:1, 1.25:1 or 0.625:1. In addition, cytokines and immunoglobulin levels measured using commercial kits as manufacturer's instruction.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Over 60 years old without any health problems
* The levels of white blood cells within range 4x10^3/μL~10x10^3/μL

Exclusion Criteria:

* Individuals who get a cold
* Diabetes
* Hypersensitivity or disease history for milk protein
* Epilepsy, neurological, or psychological disease
* Alcoholism or drug addiction
* Liver disease or severe kidney failure disease
* Inflammation-related disease
* Consumption of other test products or drugs within 1 month prior to screening
* Regular consumption of immune-related functional foods including yogurt or milk within 1 month prior to screening
* History of inflammation-related disease or taking medication to treat inflammation-related disease within 1 month prior to screening
* History of cancer within 5 years
* Any inappropriate condition

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Natural killer cell activity | At baseline
Natural killer cell activity | At 12-week follow-up
Change from baseline natural killer cell activity at 12-week | At baseline and 12-week follow-up

SECONDARY OUTCOMES:
White blood cell | At baseline
White blood cell | At 12-week follow-up
Change from baseline white blood cell at 12-week | At baseline and 12-week follow-up
Interleukin-12 | At baseline
Interleukin-12 | At 12-week follow-up
Change from baseline Interleukin-12 at 12-week | At baseline and 12-week follow-up
Interferon-gamma | At baseline
Interferon-gamma | At 12-week follow-up
Change from baseline Interferon-gamma at 12-week | At baseline and 12-week follow-up
Immunoglobulin | At baseline
Immunoglobulin | At 12-week follow-up
Change from baseline immunoglobulin at 12-week | At baseline and 12-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, Principal Investigator — Yonsei University
Locations (1):
- Yonsei University, Seoul, South Korea

REFERENCES:
- [Derived] Lee A, Lee YJ, Yoo HJ, Kim M, Chang Y, Lee DS, Lee JH. Consumption of Dairy Yogurt Containing Lactobacillus paracasei ssp. paracasei, Bifidobacterium animalis ssp. lactis and Heat-Treated Lactobacillus plantarum Improves Immune Function Including Natural Killer Cell Activity. Nutrients. 2017 May 31;9(6):558. doi: 10.3390/nu9060558. PMID 28561762